CLINICAL TRIAL: NCT00551993
Title: Conventional Laparoscopic Versus Robotic Assisted Laparoscopic Sacrocolpopexy: a Randomized Controlled Trial
Brief Title: Laparoscopic Versus Robotic Assisted Laparoscopic Sacrocolpopexy for Vaginal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-652
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: laparoscopy; robot; vaginal prolapse; sacrocolpopexy; sacral colpopexy
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Robotic Sacral Colpopexy
  Interventions: Procedure: robotic laparoscopic sacrocolpopexy
- 1 (Active Comparator): Laparoscopic Sacral Colpopexy
  Interventions: Procedure: Laparoscopic Sacral Colpopexy

INTERVENTIONS:
Procedure: robotic laparoscopic sacrocolpopexy — Da Vinci Robot
  Arms: 2
Procedure: Laparoscopic Sacral Colpopexy — Standard laparoscopy
  Arms: 1

SUMMARY:
The purpose of this study is to conduct a trial of robotic assisted versus traditional laparoscopic sacrocolpopexy in the treatment of patients with vaginal prolapse.

DETAILED DESCRIPTION:
Although laparoscopic sacrocolpopexy (LscASC) has been demonstrated to yield comparable success rates to abdominal sacrocolpopexy (93-99%) for the surgical treatment of pelvic organ prolapse, it has not been widely adopted due to the increased operating time and steep learning curves associated with laparoscopic suturing and knot-tying. For these reasons, robotic systems have been advocated for this technique. The objective of this study is to conduct a prospective single-blinded randomized controlled trial of robotic assisted versus traditional LscASC in the treatment of patients with apical vaginal prolapse stages II-IV (prolapse from 1 cm proximal to the hymen to all points distal).

This is a prospective single-blinded randomized controlled trial. Robotic assisted LscASC will be performed using the da Vinci Surgical System (Intuitive Surgical Inc., Sunnyvale, CA, USA) in a similar manner as that described above for conventional laparoscopy. Data points recorded during the procedure will include: operating room time of entry and exit, time from incision to closure and time taken for the suturing aspect of the case. From this information, the operating room costs and anesthesia costs, i.e., the amount that a provider must pay for goods or services, will be calculated. Estimated blood loss, perioperative and post-operative complications, and number of days in the hospital will be studied as will cost-effectiveness and impact on HRQOL

ELIGIBILITY:
Inclusion Criteria:

* Women who are 21 years of age or greater
* Status post hysterectomy with apical vaginal prolapse POPQ stages II-IV (prolapse from 1cm proximal to the hymen to all points distal) that desire laparoscopic surgical management.

Exclusion Criteria:

* Patients that are not candidates for general anesthesia
* Inability to consent
* History of prior sacralcolpopexy
* Suspicious adnexal masses or other factors that may indicate pelvic malignancy
* History of pelvic inflammatory disease
* Morbid obesity (body mass index greater than or equal to 40)
* History of prior or need for concomitant rectopexy with sigmoid resection.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Primary outcome: operative time from incision to closure. | Primary outcome: will be obtained immediately at the end of each procedure.

SECONDARY OUTCOMES:
Secondary outcomes: perioperative complications, hospital costs and post-operative patient outcomes (anatomic outcomes on physical examination and patient satisfaction using validated condition specific quality of life measures). | Secondary outcome: will be collected over the course of the first postoperative year

CONTACTS AND LOCATIONS:
Overall Officials: Marie Fidela M Paraiso, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Result] Paraiso MFR, Jelovsek JE, Frick A, Chen CCG, Barber MD. Laparoscopic compared with robotic sacrocolpopexy for vaginal prolapse: a randomized controlled trial. Obstet Gynecol. 2011 Nov;118(5):1005-1013. doi: 10.1097/AOG.0b013e318231537c. PMID 21979458